CLINICAL TRIAL: NCT02471807
Title: Early Feasibility Study of the Edwards FORMA Tricuspid Transcatheter Repair System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-04
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Results first posted 2022-01-06 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-02

CONDITIONS: Tricuspid Valve Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Edwards FORMA Tricuspid Transcatheter Repair System (Experimental): Edwards FORMA Tricuspid Transcatheter Repair System
  Interventions: Device: Edwards FORMA Tricuspid Transcatheter Repair System

INTERVENTIONS:
Device: Edwards FORMA Tricuspid Transcatheter Repair System

SUMMARY:
The study is a multi-center, prospective, early feasibility study to measure individual patient clinical outcomes and effectiveness, evaluate the safety and function, provide guidance for future clinical study designs and development efforts of the Edwards FORMA Tricuspid Transcatheter Repair System.

DETAILED DESCRIPTION:
The early feasibility study of the Edwards FORMA Tricuspid Transcatheter Repair System is a multi-center, prospective, early feasibility study to measure individual patient clinical outcomes and effectiveness, evaluate the safety and function, provide guidance for future clinical study designs and development efforts of the Edwards FORMA Tricuspid Transcatheter Repair System.

Data collected in this clinical study will include safety and function of the investigational system as well as up to 3 year clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. Clinically significant, symptomatic, functional, tricuspid regurgitation (per applicable guidelines) requiring transcatheter tricuspid valve repair as assessed by the local Heart Team

Exclusion Criteria:

1. Tricuspid valve/right heart anatomy not suitable for the study device
2. Moderate or greater tricuspid valve stenosis
3. Severe RV dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-12; Primary Completion 2019-06 (Actual); Study Completion 2023-01-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Emory University Hospital, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Morristown Medical Center, Morristown, New Jersey
  - Columbia University Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Edwards FORMA Tricuspid Transcatheter Repair System
Started | 34
Completed | 12
Not Completed | 22
Not completed — Death | 14
Not completed — Withdrawal by Subject | 2
Not completed — Explant | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Edwards FORMA Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 77 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (4.20)
New York Heart Association Class (NYHA) [Count of Participants; unit: Participants] — NYHA Classification -
  The stages of heart failure:
  Class I - No symptoms and no limitation in ordinary physical activity
  Class II - Mild symptoms and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than ordinary activity. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest.
  Participants
    Class I | 0
    Class II | 6
    Class III | 20
    Class IV | 8
The European System for Cardiac Operative Risk Evaluation: EuroScore II [Mean (Standard Deviation); unit: score] — The European System for Cardiac Operative Risk Evaluation (EuroSCORE II) is a risk model which allows the calculation of the risk of death after a heart operation. The higher the score, the higher the risk of an adverse outcome.
  EuroSCORE II risk levels are as follows:
  <8: Low Risk
  8-10: Moderate Risk
  >10 High Risk
  score | 7.5 (5.23)

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Event Rate : Count and Percentage of Patients Who Experienced at Least One MAE
Description: Composite of major adverse events (MAE) defined as cardiovascular mortality, myocardial infarction, new need for renal replacement therapy, severe bleeding, re-intervention for study device related complications or on the previously implanted study device, and major access site and vascular complications requiring intervention at 30 days.
Time Frame: 30 days
Population: The intention-to-treat (ITT) population includes all patients who signed informed consent, met eligibility criteria, and in whom the study procedure has been attempted (i.e. at least skin incision to introduce the FORMA System).
Measure: Count of Participants; unit: Participants
Groups:
- Edwards FORMA Tricuspid Transcatheter Repair System: Edwards FORMA Tricuspid Transcatheter Repair System Edwards FORMA Tricuspid Transcatheter Repair System
Arm/Group | Edwards FORMA Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 34
Participants | 10

2. Secondary Outcome: Device Success : Count and Percentage of Patients Who Experienced Device Success
Description: Device is deployed as intended and the delivery system is successfully retrieved as intended at the time of the patient's exit from the cardiac catheterization laboratory.
Time Frame: Intraprocedural
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards FORMA Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 34
Participants | 32

3. Secondary Outcome: Procedure Success: Count and Percentage of Patients Who Experienced Procedural Success
Description: Device success with evidence of TR reduction as evidenced by a relative reduction in EROA of ≥ 30% from baseline to discharge and without the need for a surgical or percutaneous intervention prior to hospital discharge.
Time Frame: Discharge (2-8 days)
Population: The as-treated population is a subset of ITT population and includes all patients in whom the study device is implanted and remains in position at the time of the patient's exit from the procedure room.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards FORMA Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 23
Participants | 12

4. Secondary Outcome: Clinical Success: Count and Percentage of Patients Who Experienced Clinical Success
Description: Procedural success without MAEs at 30 days. (MAEs: cardiovascular mortality, myocardial infarction, new need for renal replacement therapy, severe bleeding, re-intervention and major access site and vascular complications)
Time Frame: 30 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards FORMA Tricuspid Transcatheter Repair System
Number analyzed (Participants) | 26
Participants | 11

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Edwards FORMA Tricuspid Transcatheter Repair System
All-Cause Mortality (participants affected / at risk) | 14/34
Serious Adverse Events (participants affected / at risk) | 33/34
Other Adverse Events (participants affected / at risk) | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards FORMA Tricuspid Transcatheter Repair System (N=34)
Anaemia (Blood and lymphatic system disorders) | 7 (7)
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1)
Ascites (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3)
Cardiac failure (Cardiac disorders) | 13 (23)
Cardiac failure acute (Cardiac disorders) | 3 (4)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2)
Dyspnoea (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (7)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 3 (3)
Device related thrombosis (General disorders) | 1 (1)
General disorders and administration site conditions (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Ulcer haemorrhage (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic encephalopathy (Hepatobiliary disorders) | 2 (3)
Cellulitis (Infections and infestations) | 2 (2)
Endocarditis staphylococcal (Infections and infestations) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (4)
Klebsiella infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Pneumonia serratia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Application site wound (Injury, poisoning and procedural complications) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Cardiac perforation (Injury, poisoning and procedural complications) | 2 (2)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
International normalised ratio increase (Investigations) | 2 (2)
Occult blood positive (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Constochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Device dislocation (Product Issues) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Renal failure (Renal and urinary disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 (1)
Glaucoma surgery (Surgical and medical procedures) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Epistaxis (Vascular disorders) | 1 (2)
Gastrointestinal haemorrhage (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (4)
Internal haemorrhage (Vascular disorders) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1)
Rectal haemorrhage (Vascular disorders) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 1 (1)
Post procedural hypotention (Injury, poisoning and procedural complications) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards FORMA Tricuspid Transcatheter Repair System (N=34)
Anaemia (Blood and lymphatic system disorders) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Ascites (Cardiac disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Bundle branch block right (Cardiac disorders) | 3 (3)
Cardiac failure (Cardiac disorders) | 6 (6)
Pericardial effusion (Cardiac disorders) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Myocardial necrosis marker increased (Investigations) | 2 (2)
Troponin increased (Investigations) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 3 (4)
Haematuria (Renal and urinary disorders) | 2 (3)
Urinary retention (Renal and urinary disorders) | 4 (5)
Hypotension (Vascular disorders) | 4 (4)
Renal failure (Renal and urinary disorders) | 6 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Genitourinary tract infections and inflammation NEC (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol: Rev K (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT02471807/Prot_000.pdf
  • Study Protocol: Rev M (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT02471807/Prot_001.pdf
  • Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT02471807/SAP_002.pdf